CLINICAL TRIAL: NCT06505174
Title: Effect of Treatment With Systane Ultra in Symptomatology and Visual Task Efficiency in Digital Device Users
Status: Completed | Type: Observational
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Raul Martin Herranz, PhD, University of Valladolid
Other Study IDs: UVaGiO-PI222911
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Digital Eye Strain; Computer Vision Syndrome; OSDI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Use of hydroxypropyl Guar-based artificial tears four times per day: Use of hydroxypropyl Guar-based artificial tears four times per day
  Interventions: Other: Hydroxypropyl Guar-based artificial tears four times per day

INTERVENTIONS:
Other: Hydroxypropyl Guar-based artificial tears four times per day — Use of hydroxypropyl Guar-based artificial tears four times per day

SUMMARY:
This study assessed the effect of one month of use of preservative-free artificial tears (Systane Ultra UD, Alcon) on symptomatology related to digital eye strain (DES), visual task performance, and tear film stability in visual display terminal users.

DETAILED DESCRIPTION:
Visual display terminal users (>4h/day) with DES (CVSS17 score: ranged 29 to 42) and dryness (OSDI score: ranged 13 to 24) symptomatology were prescribed with preservative-free artificial tears (Systane Ultra UD, Alcon) four times a day for one month collecting OSDI and CVSS17 questionnaires in four visits [screening (Day -7), initial (Day 0), one week (Day 7) and one month (Day 30)].

Blink rate and number of eye fixations (collected with eye-tracker) in six simple computer tasks and out-loud reading speed were determined before and after performing all tasks on the computer. Tear film stability and ocular parameters were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subjects of legal age will be included who agree to participate in the study after being informed by the researcher, receiving the information sheet and signing the informed consent.
* Eye discomfort related to dryness (OSDI score ranged from 13 to 24)
* Symptomatic digital device users (CVSS17 score ranged from 29 to 42 points - stages 3 and 4)
* Use of computer continuously for at least 4 hours per day (work week)
* Good best-corrected visual acuity (Visual acuity LogMar ≤ 0.00 for distance, intermediate (60cm) and near (40cm))

Exclusion Criteria:

* Systemic administration of drugs with a possible effect on the ocular surface.
* Topical administration of any drugs that can alter the ocular surface.
* Use of contact lenses
* Use of artificial tears or lubricants at least 7 days before inclusion in the study (recruitment visit).
* Any other ocular pathology or binocular conditions which may cause discomfort (e.g. heterophoric, accommodative, and eye movement disorders)

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
OSDI Score | One month
  Change in OSDI score
CVSS17 Score | One month
  Change in CVSS17 score

CONTACTS AND LOCATIONS:
Locations (1):
- IOBA Eye Institute, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be available by reasonable request to PI